CLINICAL TRIAL: NCT05277935
Title: Wearable Enhanced Fitness Tracking for Metastatic Breast Cancer Patients Using Endocrine Treatment and Palbociclib
Acronym: WEFITTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beneficência Portuguesa de São Paulo (Other)
Responsible Party: Principal Investigator, Graziela Zibetti Dal Molin, MD, Beneficência Portuguesa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: WEFITTER
Record Dates: First submitted 2022-01-12; First posted 2022-03-14 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Breast Neoplasm Female; Quality of Life
Keywords: Quality of life; Metastatic breast cancer; Metastasis; Exercise; Palbociclib
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of the WeCancer app combined with the smartwatch (Active Comparator): The Wecancer app will be used in a way, combined with a smartwatch, similar to those used in professional fitness programs, with active measures, which may include, for example: notifications with personalized advice (via chat), feedback to the patient in the comments made, guidance on physical and eating exercises, reception and support from the Wecancer multidisciplinary team, consisting of a navigator nurse, psychologist, nutritionist and physiotherapist. During the survey period, participants should report their symptoms on the Wecancer app whenever possible, preferably daily.
  Interventions: Device: Use of the WeCancer app combined with the smartwatch.
- Using the WeCancer app (No Intervention): The Wecancer application similar to those used in professional fitness programs, with active measures, which may include, for example: notifications with personalized advice (via chat), patient feedback on the comments made, guidance on physical and dietary exercises, reception and support of the Multidisciplinary cancer team composed of a navigator nurse, a psychologist, nutritionist and physiotherapist. During the research period, participants must report your symptoms in the Wecancer app whenever possible, preferably daily.

INTERVENTIONS:
Device: Use of the WeCancer app combined with the smartwatch. — To evaluate if a fitness tracker added to eHealth technology will improve quality of life compared to the use of eHealth technology alone in metastasis breast cancer patients treated with palbociclib and endocrine therapy
  Arms: Use of the WeCancer app combined with the smartwatch

SUMMARY:
Combining a fitness tracker technology with real-time patient-reported outcome monitoring associated with interventions through a health care app is a novel strategy to evaluate metastatic breast cancer patients using Palbociclib and endocrine treatment.

DETAILED DESCRIPTION:
Measure the quality of life of patients with metastatic breast cancer treated with Palbociclib and endocrine therapy using the Functional Assessment of Cancer Therapy - Breast and EuroQol -5D - European quality of life in five dimensions and compare the group using the Wecancer digital health app with the group using Wecancer and the physical activity monitoring smartwatch.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥ 18 years of age diagnosed with hormone receptor-positive/ human epidermal growth factor receptor 2- negative metastatic breast cancer undergoing treatment with Palbociclib combined with aromatase inhibitors (letrozole, exemestane or anastrozole) or fulvestrant as first-line therapy, or in treatment with Palbociclib and fulvestrant as second-line or posterior-line therapy in the metastatic setting; may be using ovarian suppression if the patient is premenopausal.
* The patient must be on treatment for at least three (3) months with Palbociclib and endocrine therapy.
* Evidence of a signed and dated informed consent document, physically or digitally, indicating that the research participant was informed about all relevant aspects of the study;
* The patient agrees not to participate in another study with drug intervention while on treatment.
* Have performance status according to the Eastern Cooperative Oncology Group
* Have access to a compatible smartphone and 3G or 4G internet connection

Exclusion Criteria:

* Patients considered to be at poor medical risk due to uncontrolled serious medical disorder, non-malignant systemic disease, or active uncontrolled infection. Examples: uncontrolled ventricular arrhythmia, recent myocardial infarction (within 6 months), stroke, gastrointestinal bleeding, or any psychiatric disorder that precludes informed consent; between others.
* Patients who have a life expectancy of < 3 months.
* Treatment with any product under investigation during the last 28 days;
* Another acute or chronic medical or psychiatric condition or severe laboratory abnormality that could increase the risk associated with participation in the study or that Page 10 de 21 Version 6.0 could interfere with the interpretation of the study results and, in the investigator's judgment, would make the research participant unsuitable for inclusion in the study. study.
* Illiterate patients or those with a low level of education that may prevent the correct use of the Wecancer application and/or the watch with monitoring of physical activity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Assess quality of life through the quality-of-life questionnaire through the Functional Assessment of Cancer Therapy - Breast | Baseline
  Measure the Quality of life of patients with metastatic breast cancer treated with Palbociclib and endocrine therapy using the Functional Assessment of Cancer Therapy - Breast and compare the group using the Wecancer digital health app with the group using Wecancer and the physical activity monitoring smartwatch.
  The comparison of the two groups in relation to quality of life, measured by the general score of the Functional Assessment of Cancer Therapy - Breast and its sub-items, over time will be made using a linear model withmixed effects, that is, fixed effects and random effects. Time and group fixed effects will be considered, the patient will be considered random effect. The effects of time, group and interaction between them will be tested.
Assess quality of life through the quality-of-life questionnaire through the Functional Assessment of Cancer Therapy - Breast | Follow up 2 month
  Measure the Quality of life of patients with metastatic breast cancer treated with Palbociclib and endocrine therapy using the Functional Assessment of Cancer Therapy - Breast and compare the group using the Wecancer digital health app with the group using Wecancer and the physical activity monitoring smartwatch.
  The comparison of the two groups in relation to quality of life, measured by the general score of the Functional Assessment of Cancer Therapy - Breast and its sub-items, over time will be made using a linear model withmixed effects, that is, fixed effects and random effects. Time and group fixed effects will be considered, the patient will be considered random effect. The effects of time, group and interaction between them will be tested.
Assess quality of life through the quality-of-life questionnaire through the Functional Assessment of Cancer Therapy - Breast | Follow up 4 month
  Measure the Quality of life of patients with metastatic breast cancer treated with Palbociclib and endocrine therapy using the Functional Assessment of Cancer Therapy - Breast and compare the group using the Wecancer digital health app with the group using Wecancer and the physical activity monitoring smartwatch.
  The comparison of the two groups in relation to quality of life, measured by the general score of the Functional Assessment of Cancer Therapy - Breast and its sub-items, over time will be made using a linear model withmixed effects, that is, fixed effects and random effects. Time and group fixed effects will be considered, the patient will be considered random effect. The effects of time, group and interaction between them will be tested.
Assess quality of life through the quality-of-life questionnaire through the Functional Assessment of Cancer Therapy - Breast | Follow up 6 month
  Measure the Quality of life of patients with metastatic breast cancer treated with Palbociclib and endocrine therapy using the Functional Assessment of Cancer Therapy - Breast and compare the group using the Wecancer digital health app with the group using Wecancer and the physical activity monitoring smartwatch.
  The comparison of the two groups in relation to quality of life, measured by the general score of the Functional Assessment of Cancer Therapy - Breast and its sub-items, over time will be made using a linear model withmixed effects, that is, fixed effects and random effects. Time and group fixed effects will be considered, the patient will be considered random effect. The effects of time, group and interaction between them will be tested.

CONTACTS AND LOCATIONS:
Overall Officials: Graziela Dal Molin, MD, Principal Investigator — Beneficência Portuguesa de São Paulo
Locations (4):
- Brazil (4):
  - Oncoclínicas, Rio de Janeiro
  - A Beneficência Portuguesa de São Paulo, São Paulo
  - A.C.Camargo Cancer Center, São Paulo
  - Centro Paulista de Oncologia, São Paulo